CLINICAL TRIAL: NCT01543113
Title: cKIT, BRAF/NRAS Mutations in Advanced Melanoma : Clinical Outcome in Response to Tyrosine-kinase Inhibitors - KitMel Project
Acronym: KitMel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOC/10-16 - KitMel; 2010-A01310-39 (Other: AFSSAPS); 10/43-785 (Other: CPP Ouest V (Rennes)); 11.272 (Other: CCTIRS); 911305 (Other: CNIL)
Record Dates: First submitted 2012-02-21; First posted 2012-03-02 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Melanoma
Keywords: melanoma; white-caucasian population
MeSH Terms: conditions — Melanoma | interventions — Base Sequence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- melanoma (Other): melanoma
  Interventions: Other: sequencing

INTERVENTIONS:
Other: sequencing — sequencing

SUMMARY:
Background: Metastatic melanoma has a devastating prognosis and is one of the top causes of cancer death in young patients. Until now, available therapies were few and unreliable, but recent understanding of melanomas' molecular pathways has improve their classification and new clinical strategies have been proposed.

Initial studies showed that B-Raf/N-Ras mutations (respectively V600E and Q61) are the most frequent alteration being present in 70 to 80% of melanomas, characterizing non Chronic Sun-induced Damage skins (CSD). These include Superficial Spreading Melanomas (SSM) and Nodular Melanomas (NM). Other studies showed that c-Kit mutations are presently the predominant activating mutation (20 - 40 %) in Acro-Lentiginous Melanomas (ALM), Mucous Melanomas (MM) and in melanomas arising on CSD skin. c-Kit mutation pattern is more complex with four exons being affected leading to different mutations, which incidence and biological impact are less documented.

BRAF/NRAS genetics alterations drive constantly cell growth, being thus attractive targets. Spectacular results have indeed been obtained with the BRAF inhibitor that targets the V600E BRAF-mutated form. Data from GIST disease revealed that the different c-Kit mutations modulate differently c-Kit function and the response to targeted therapies.

Because c-Kit targeted therapy is a critical clinical issue, the investigators aimed to identify the most frequent mutations present in our population to propose appropriate screening test and adapt the therapy.

Methods: 250 melanoma samples corresponding to an homogeneous white-Caucasian population (Brittany, France) will be screened. c-Kit exons 11, 13, 17 and 18 will be sequenced (direct sequencing and pyrosequencing when possible). c-Kit copy number will be quantified by q-PCR and level of c-Kit determined by immunohistochemistry (IHC, CD117). Samples will also be analyzed for B-Raf mutations in codon 464, 466, 469 and 600, and for N-Ras mutations in codon 12, 13 and 61 (Pyrosequencing).

Expected Results:

Taken together, the investigators anticipate that the present genetic analysis of the tumours from patients with advanced melanoma will first document the type and frequency of cKit mutations, will confirm or not that BRAF, NRAS and cKit mutations are mutually exclusive and document their repartition in the melanomas sub-types. Finally this study will clue researchers in to how well patients will respond to a therapy that targets the growth-promoting proteins BRAF/NRAS and cKIT.

ELIGIBILITY:
Inclusion Criteria:

* melanoma
* white caucasian population

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
c-Kit exons 11, 13, 17 and 18 will be sequenced (direct sequencing and pyrosequencing when possible) | Day 1
  c-Kit exons 11, 13, 17 and 18 will be sequenced (direct sequencing and pyrosequencing when possible)

SECONDARY OUTCOMES:
level of c-Kit determined by immunohistochemistry | Day 1
  level of c-Kit determined by immunohistochemistry
Samples will also be analyzed for B-Raf mutations in codon 464, 466, 469 and 600, and for N-Ras mutations in codon 12, 13 and 61 (Pyrosequencing). | Day 1
  Samples will also be analyzed for B-Raf mutations in codon 464, 466, 469 and 600, and for N-Ras mutations in codon 12, 13 and 61 (Pyrosequencing).

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Dominique Galibert, PU-PH, Principal Investigator — Rennes University Hospital
Locations (2):
- France (2):
  - Centre Eugène Marquis, Rennes, Brittany Region
  - Rennes University Hospital, Rennes, Brittany Region

REFERENCES:
- [Result] Pracht M, Mogha A, Lespagnol A, Fautrel A, Mouchet N, Le Gall F, Paumier V, Lefeuvre-Plesse C, Rioux-Leclerc N, Mosser J, Oger E, Adamski H, Galibert MD, Lesimple T. Prognostic and predictive values of oncogenic BRAF, NRAS, c-KIT and MITF in cutaneous and mucous melanoma. J Eur Acad Dermatol Venereol. 2015 Aug;29(8):1530-8. doi: 10.1111/jdv.12910. Epub 2015 Jan 26. PMID 25623140